CLINICAL TRIAL: NCT03774121
Title: Cryoneurolysis for the Management of Chronic Pain in Patients With Knee Osteoarthritis; A Randomized Controlled Study
Brief Title: Cryoneurolysis for the Management of Chronic Pain in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Niels-Peter Brøchner Nielsen, PhD, Post doc, Research employee, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CryoKnee01
Record Dates: First submitted 2018-12-03; First posted 2018-12-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain; Osteoarthritis, Knee
Keywords: Cryoneurolysis; Exercise; Pain; Physical capacity
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee; Motor Activity; Pain | interventions — Cryosurgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRYO (Experimental): Subjected to Cryoneurolysis treatment and Neuromuscular training (GLA:D).
  Interventions: Device: Cryoneurolysis; Other: Neuromuscular exercise (GLA:D)
- SHAM (Sham Comparator): Subjected to similar procedures as CRYO, but without freezing temperatures. Subjected to Neuromuscular training (GLA:D).
  Interventions: Other: Neuromuscular exercise (GLA:D); Device: Sham

INTERVENTIONS:
Device: Cryoneurolysis — A cryoprobe will be inserted percutaneously and freeze the target nerves (infrapatellar branch of the saphenous nerve & anterior femoral cutaneous nerve) guided by ultrasound visualization.
  Other Names: Cryoablation
  Arms: CRYO
Other: Neuromuscular exercise (GLA:D) — The GLA:D program, is a standard education and exercise program for patients with osteoarthritis in Denmark. The program is performed in groups and with the supervision of an experienced physiotherapist specialized in training of musculoskeletal disorders.
Device: Sham — The sham intervention includes a similar procedure but without freezing temperatures.
  Arms: SHAM

SUMMARY:
Pain is the principal symptom in knee osteoarthritis (OA) and results in a considerable amount of years lived with disability, emotional distress and has significant socioeconomic consequences. Conservative treatment options, such as exercise, often fail to provide long-term pain relief and alternatively patients may be subjected to total knee arthroplasty. More than 20% of these patients experience persistent and unchanged pain post-surgery. Novel advances in the field of cryoneurolysis applies low temperatures to disrupt nerve signaling at the painful area and a recent study showed that it was possible to target the peripheral nerves in the knee and provide significant pain relief in patients with knee OA. This could potentially improve the efficacy of other therapies such as exercise, delaying or perhaps avoiding surgical intervention and improving quality of life in OA patients considerably. Further prospective randomized controlled studies are needed to confirm the effects of cryoneurolysis treatment in patients with knee OA. The primary objective of the current project is to determine the effectiveness of cryoneurolysis in its ability to decrease pain in patients with knee OA. The secondary objective is to evaluate the safety and effectiveness of cryoneurolysis in its ability to improve outcomes in the GLA:D program to potentially delay or avoid surgical intervention. 90 individuals with knee OA in the knee will be randomly allocated in either a cryoneurolysis intervention group or a sham group. Both groups will be assessed at baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up. The patients, therapists and data-manager will be blinded to the allocation. The primary outcome will be VAS knee pain intensity score, measured post cryoneurolysis treatment. Secondary outcome measures include functional performance, PRO-data (KOOS, EQ5D), analgesic use, a socio-economic evaluation and adverse effects.

DETAILED DESCRIPTION:
BACKGROUND Pain is the principal symptom in knee osteoarthritis (OA) and results in a considerable amount of years lived with disability, emotional distress and has significant socioeconomic consequences. Knee OA in particular, has a high prevalence rate compared to other types of OA, and is also present in the younger working age population. The treatment of knee OA typically focuses on pain relief, however the effects of current conservative treatment options remain small to moderate and most are associated with side effects. In many cases patients alternatively may be subjected to partial/total knee arthroplasty (TKA). TKA is considered to be an effective treatment for end-stage knee osteoarthritis however more than 20% of patients receiving TKA, experience persistent and unchanged pain post-surgery. Reviewing these results, focus should be on low-risk, minimally invasive therapies. Novel advances in the field of cryoneurolysis are in that respect promising. Cryoneurolysis has made it possible to apply low temperatures to a target percutaneous peripheral nerve, causing Wallerian degeneration. This has been shown to provide pain relief in a variety of chronic pain conditions. Recently, Radnovich et al. (2017) targeted the genicular nerves to reduce pain in patients with knee OA. The authors reported significant pain relief in patients with knee OA for up to 150 days. The authors reported expected adverse effects, that were transient, with mild severity, requiring no further intervention. These results might suggest that cryoneurolysis treatment is a safe procedure, that may reduce both pain and symptoms in patients with knee OA. Further prospective randomized controlled studies, with adequate power are needed to confirm the efficacy and safety of cryoneurolysis treatment in patients with knee OA.

In Denmark, a neuromuscular exercise program (GLA:D) has been implemented, for the treatment of knee and hip OA in clinical practice. Recent studies show that exercise reduce pain and improve function in people with knee or hip OA. Despite of these reports the beneficial effects remains moderate with difficulties in maintaining these effects at long-term follow-up and includes a significant discontinuation rate for patients reporting high pain levels. In this line, pain and muscle weakness, among others, have been reported to be major barriers for physical exercise. The application of cryoneurolysis treatment as an effective pain reducing treatment prior to a standardized exercise program could perhaps provide significant pain relief, resulting in improved adherence, exercise effectiveness and long-term benefits of both therapies.

The primary objective of the current project is to determine the effectiveness of cryoneurolysis in its proposed ability to decrease pain in patients with knee osteoarthritis. The secondary objective is to evaluate the safety and effectiveness of cryoneurolysis in its ability to improve outcomes in the GLA:D program to potentially delay or avoid surgical intervention.

We hypothesize that cryoneurolysis in combination with GLA:D will be a safe and effective therapeutic option with few side effects to reduce pain in patients with knee osteoarthritis and may post pone surgical intervention.

TRIAL DESIGN This study is a randomized, controlled, trial (RCT) designed to test the efficacy of cryoneurolysis treatment in patients with knee osteoarthritis followed by a neuromuscular exercise program (GLA:D). The patients will be randomly allocated in either a cryoneurolysis intervention group (CRYO) or a sham group (SHAM) and will be assessed at baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up. The tests will include both patient-reported outcomes (PRO) and objective functional measurements.

RECRUITMENT AND SAMPLE SIZE Patients with pain and knee OA confirmed by radiography, are referred to GLA:D by their general practitioner prior to assessment of surgery eligibility at the hospital. The current project will recruit these patients in collaboration with selected general practitioners in the Region of Southern Denmark. According the Region of Southern Denmark, an average of 270 patients participate in the GLA:D program every year. Based on this estimation and considering the eligibility criteria to participate in the current project, recruitment will continue for up to 1 year.

The planned number of trial participants is based on the assumed superiority of the cryoneurolysis treatment over control. Estimating the sample size for a two-sample means test with a level of significance at 0.05, assuming a common standard deviation (SD) of 30 in VAS pain intensity scores indicates that for the intention-to-treat (ITT) population, 74 individuals is required to obtain a power of at least 80% to establish a minimal clinically significant difference (MCSD) of 20 in VAS pain scores. The MCSD and common standard deviation is based on previous findings with a similar patient group and intervention. With an expected drop-out rate of 20%, a total of 94 individuals will be included in the project, 47 in each group.

ALLOCATION AND BLINDING Randomization will be performed as computer-generated block randomization with a 1:1 allocation ratio using random block sizes of 2, 4 and 6 in either group CRYO or group SHAM. The randomization restrictions will not be disclosed to ensure allocation concealment and the sequence will be performed by an external co-investigator.

To account for the placebo effect and reduce the risk of bias, the patients, therapists and data-manager will be blinded to the allocation. Blinding will be assured using a sham trial that includes the same procedures as cryoneurolysis treatment but without any freezing temperatures. Thus, visible marks as a result of the procedures in both groups will be similar.

INTERVENTIONS Diagnostic nerve block. All patients reporting a decrease of ≥ 50 % in VAS pain scores at least 15 min after a diagnostic nerve block of the genicular nerves.

Cryoneurolysis. The current project involves the novel application and test of cryoneurolysis, in the treatment of OA related pain. The rationale behind this method, is based on previous reports showing that low temperature conditions can alter nerve function. This technology allows for reversible destruction of nerves, also known as Wallerian degeneration, that prevents nerve signaling and potentially alleviate pain and motor dysfunction in a number of medical conditions. A probe will be inserted percutaneously at the target anterior femoral cutaneous nerve and infrapatellar branch of the saphenous nerve guided by ultrasound visualization to accurately determine the location of the nerve and to account for adjacent neurovascular structures and variations in anatomical structures. The target locations are drawn directly on the patients' skin prior to treatment along which a dose of local anesthetic will be injected subcutaneously before treatment. Cryoneurolysis at each target site requires 2-4 freeze cycles with a duration of 3 mins, and with thaw cycles between 20-40 seconds. A temperature probe will be inserted adjacent to the target nerve and cryoneurolysis-probe to ensure a controlled cooling effect and to control nerve damage. The sham intervention includes a similar procedure but using a sham probe.

GLA:D. SHAM and CRYO will both participate in the GLA:D program, which is a standard education and exercise program for patients with osteoarthritis in Denmark. The program is performed in groups and with the supervision of an experienced physiotherapist specialized in training of musculoskeletal disorders and has a duration of 8 weeks.

STATISTICAL METHODS The treatment groups will be examined for comparability based on baseline demographic and prognostic measures. An Intention-To-Treat (ITT) analysis will be used for all allocated patients and a mixed effects model will be used on the continuous outcome measures to determine the effects of cryoneurolysis treatment from baseline to post treatment and follow-ups [Between groups factor: CRYO vs SHAM, within groups factor: time]. The model will use robust estimation methods to account for outliers. Finally, a multiple imputation approach will be used in case of missing data. All P-values < 0.05 will be considered statistically significant.

ETHICS AND SIGNIFICANCE The project will be conducted according to the declaration of Helsinki and will be registered in ClinicalTrials.gov. The Project has been approved by the Regional Committee on Health Research Ethics for Southern Denmark (S-20180089).

Cryoneurolysis could potentially provide an effective, safe and minimally invasive option to treat pain in OA patients. The potential benefits include increased functional capacity and quality of life as a result of significant pain relief and improved benefits of physical exercise, ultimately postponing or making surgical intervention unnecessary. Finally, an important perspective, is the application of cryoneurolysis in other areas - such as managing pain, related to surgery, to improve rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Referred to GLA:D by a physician.
* Age ≥ 18y
* Chronic knee pain for a minimum duration of 6 months.
* Pain intensity ≥ 40mm on a 100mm visual analogue scale (VAS).
* Radiographic confirmation of osteoarthritis; Grade 2-4 changes according to the Kellgren Lawrence classification system
* A decrease of ≥ 50 % in VAS scores with diagnostic genicular nerve block.
* Written and oral understanding of Danish.

Exclusion Criteria:

* History of systemic inflammatory conditions such as rheumatoid arthritis.
* Previous recipient of cryoneurolysis for the knee.
* Use of hyaluronic acid within the previous 30 days.
* Injection of corticosteroid within the previous 3 months.
* Clinical significant structural abnormities affecting locomotion and knee function aside from osteoarthritis and which might cause chronic knee pain.
* Body mass index ≥ 18 and ≤ 40 kg/m
* In treatment for other pain conditions.
* Pregnancy
* Coagulopathy
* Uncontrolled serious disease (cancer, diabetes, etc.)
* Disease associated with reactions to cold, such as cryoglobulinemia, cold urticarial and Renaud's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in NRS knee pain intensity score | Change in NRS pain score, between baseline and two weeks post surgery
  NRS consists of a numerical, from 0 to 10, anchored by two verbal descriptors, "no pain" for the score of zero and "worst pain imaginable" for the score of 10. NRS is a self-reported tool where the respondent is asked their current pain intensity.

SECONDARY OUTCOMES:
Change in Pain location | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  Pain location as drawn by the patient.
Change in Functional Performance Evaluated by the 30 second chair-stand test. | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  The outcome is the total number of complete chair stands performed for the duration of the task (one chair stand represents a stand followed by a sit movement).
Change in use of Analgesics | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  Use of analgesics from medical records
Number of Adverse effects | Reported adverse effects 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  Pre-defined and unexpected adverse effects
Change in Pain type | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  Change in pain type using prespecified pain definitions
Change in Functional Performance Evaluated by the 40m fast-paced walk test. | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  The outcome is expressed as speed. i.e. walking distance (40m) divided by the time to perform the task (s).
Change in Functional Performance Evaluated by the 9 step stair test. | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  The outcome is the total time to perform the task (s).
Change in Functional Performance Evaluated by Maximum Voluntary Contraction | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  As measured in moment force of the knee extensors (Nm)
Change in Quality of Life using the Quality of Life questionnaire (EQ5D) | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  EQ5D consists of 5 subscales; Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety / depression. An health state score is obtained based on the responses from 1-5 in each subscale, from which a single index value is calculated representing patients' overall health state.
Change in self-rated health using the Quality of Life questionnaire (EQ5D) | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  EQ5D includes a so called EQ VAS score which is the patients' self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled "the best health you can imagine" and "the worst health you can imagine".
Change in the subscale "Pain" using the Knee injury and Osteoarthritis Score (KOOS score) | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) us calculated for each subscale.
Change in the subscale "other Symptoms" using the Knee injury and Osteoarthritis Score (KOOS score) | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) us calculated for each subscale.
Change in the subscale "Function in daily living (ADL)" using the Knee injury and Osteoarthritis Score (KOOS score) | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) us calculated for each subscale.
Change in the subscale "Function in sport and recreation (Sport/Rec)" using the Knee injury and Osteoarthritis Score (KOOS score) | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) us calculated for each subscale.
Change in the subscale "Knee related Quality of Life (QoL)" using the Knee injury and Osteoarthritis Score (KOOS score) | Change between baseline, 2 weeks post cryoneurolysis, post GLA;D and at 6, 12 and 24 month follow-up.
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) us calculated for each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Bibi (Valgerdur) Gram, PhD, Study Director — Esbjerg Hospital - University Hospital of Southern Denmark; Carsten Kock-Jensen, MD, Study Director — Esbjerg Hospital - University Hospital of Southern Denmark; Niels-Peter B Nielsen, PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of Southwest Jutland, Esbjerg, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] SUNDERLAND S. A classification of peripheral nerve injuries producing loss of function. Brain. 1951 Dec;74(4):491-516. doi: 10.1093/brain/74.4.491. No abstract available. PMID 14895767
- [Background] Ilfeld BM, Preciado J, Trescot AM. Novel cryoneurolysis device for the treatment of sensory and motor peripheral nerves. Expert Rev Med Devices. 2016 Aug;13(8):713-25. doi: 10.1080/17434440.2016.1204229. Epub 2016 Jul 13. PMID 27333989
- [Background] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454
- [Background] Trescot AM. Cryoanalgesia in interventional pain management. Pain Physician. 2003 Jul;6(3):345-60. PMID 16880882
- [Background] Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D): evidence-based education and supervised neuromuscular exercise delivered by certified physiotherapists nationwide. BMC Musculoskelet Disord. 2017 Feb 7;18(1):72. doi: 10.1186/s12891-017-1439-y. PMID 28173795
- [Background] Dasa V, Lensing G, Parsons M, Harris J, Volaufova J, Bliss R. Percutaneous freezing of sensory nerves prior to total knee arthroplasty. Knee. 2016 Jun;23(3):523-8. doi: 10.1016/j.knee.2016.01.011. Epub 2016 Feb 10. PMID 26875052
- [Background] Lewis GN, Rice DA, McNair PJ, Kluger M. Predictors of persistent pain after total knee arthroplasty: a systematic review and meta-analysis. Br J Anaesth. 2015 Apr;114(4):551-61. doi: 10.1093/bja/aeu441. Epub 2014 Dec 26. PMID 25542191
- [Background] O'Brien T, Breivik H. The impact of chronic pain-European patients' perspective over 12 months. Scand J Pain. 2012 Jan 1;3(1):23-29. doi: 10.1016/j.sjpain.2011.11.004. PMID 29913762
- [Background] Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. BMC Musculoskelet Disord. 2010 Jun 17;11:126. doi: 10.1186/1471-2474-11-126. PMID 20565735
- [Derived] Nygaard NB, Koch-Jensen C, Vaegter HB, Wedderkopp N, Blichfeldt-Eckhardt M, Gram B. Cryoneurolysis for the management of chronic pain in patients with knee osteoarthritis; a double-blinded randomized controlled sham trial. BMC Musculoskelet Disord. 2021 Feb 26;22(1):228. doi: 10.1186/s12891-021-04102-1. PMID 33637085

DOCUMENTS (2):
  • Study Protocol (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT03774121/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT03774121/SAP_001.pdf